CLINICAL TRIAL: NCT05960539
Title: Robotic Curriculum for Young Surgeons
Acronym: RoCS
Status: Recruiting | Type: Observational
Sponsor: Otto-von-Guericke University Magdeburg (Other)
Responsible Party: Principal Investigator, Jessica Stockheim, MD, Otto-von-Guericke University Magdeburg
Other Study IDs: 152/20
Record Dates: First submitted 2022-02-20; First posted 2023-07-25 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Robotic Surgery
Keywords: robotic surgery; NASA Task Load Index; training; curriculum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- robotic procedures: surgical residents and experts; differentiation due to organ systems
  Interventions: Procedure: surgical training

INTERVENTIONS:
Procedure: surgical training — surgical residency focussed on visceral robotic procedures

SUMMARY:
Robotic training program for unexperienced novice surgeons

DETAILED DESCRIPTION:
The curricular structure of RoCS bases on five modules: multimodular didactics, standardization, training structure, interdisciplinary workplace and evaluation. The aim is to ensure a basic competence of robotic surgcial skills for unexperienced novice surgeons (residents).

ELIGIBILITY:
Inclusion Criteria:

* robotic procedures

Exclusion Criteria:

* no consent of patients or surgeons

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * every surgery for which patients gave their consent to participating in the study
  * every surgeon giving consent of collecting data via this study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
perioperative morbidity | 5 years
  complications classified by Clavien-Dindo
patient mortality rate | 5 years
  during in-hospital stay, 30 and 90 days postoperatively
intraoperative workload | 5 years
  The questionnaire NASA Task Load Index consists of 6 quesions addressing the individual overall workload. The question of level of procedure's difficulty is used to analyse the overall workload additionally referring to "Lowndes BR, Forsyth KL, Blocker RC, Dean PG, Truty MJ, Heller SF, Blackmon S, Hallbeck MS, Nelson H. NASA-TLX Assessment of Surgeon Workload Variation Across Specialties. Ann Surg. 2020 Apr;271(4):686-692. doi: 10.1097/SLA.0000000000003058. PMID: 30247331."
basic robotic competence | 5 years
  Evaluation of the intraoperative performance of residents and specialists by the robotic expert using O-SCORE referring to doi:10.1097/ACM.0b013e3182677805. PMID: 22914526

SECONDARY OUTCOMES:
patient characteristics | 5 years
  age, sex, BMI, preexisting illnesses and diseases
patient laboratory parameters | 5 years
  pre- and postoperatively: concentration of hemoglobin and tsh, crp value, estimated glomerular filtration rate, concentration of albumin, prothrombin time
surgical expertise | 5 years
  analysis of experience for open, laparoscopic and robotic procedures by counting numbers of procedures and surgical practice in years
practical resident training | 5 years
  percentage of intraoperative procedural steps performed by the assisting surgeon
robotic bedside assistance | 5 years
  analysis of duration of port placement and docking in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Roland S. Croner, Prof., Study Director — Otto-von-Guericke University of Magdeburg
Locations (1):
- Otto-von-Guericke University Magdeburg, Magdeburg, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: Undecided